CLINICAL TRIAL: NCT03520608
Title: Painful Diabetic Peripheral Neuropathy Study of Chinese OutPatiEnt (PDN-SCOPE): a Multi-center Cross-sectional Registry Study of Clinical Characteristics and Treatment Survey of PDN in China
Brief Title: Painful Diabetic Peripheral Neuropathy Study of Chinese OutPatiEnt
Acronym: SCOPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Fan Dongsheng, Director, Peking University Third Hospital, Neurology Depatment, Peking University Third Hospital
Other Study IDs: 2018182
Record Dates: First submitted 2018-04-09; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Painful Diabetic Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Painful Diabetic peripheral Neuropathy Study of Chinese OutPatiEnt (PDN-SCOPE): a multi-center cross-sectional registry study of clinical characteristics and treatment survey of PDN in China

DETAILED DESCRIPTION:
Painful diabetic peripheral neuropathy (PDN) presents a serious health problem in China. SCOPE is a cross-sectional, multi-centers registry study with a target sample size of 1500 patients who are experiencing PDN. The patients are treated following guideline and local practice. Real-world data including demographics, medical histories, VAS, PHQ, GAD -7 and therapies are collected. The primary objective is to analyze the clinical characteristics of PDN. The secondary objectives include anxiety depression distribution and current treatment status.The SCOPE study will help to find actual clinical manifestation and treatment and improve the overall treatment outcome of Chinese patients with PDN.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older patients
2. definite diagnosis of type I and type II diabetes
3. evidence of symptoms, signs and/or electrophysiology of diabetic peripheral neuropathy
4. complains of spontaneous pain (continuous or intermittent needle pricking, electric pain, burning pain etc.) or induced pain (hypersensitivity, sensory inversion).
5. the pain lasts for at least 3 months
6. signed informed consent

Exclusion Criteria:

1. other causes of neuropathic pain, non-neuropathic pain or mixed pain, such as neck / lumbar degenerative disease, arthritis, nerve root compression, para-neoplastic syndrome, cerebrovascular disease, spinal cord diseases and other peripheral neuropathy (immunity, toxic and nutritional neuropathy etc.)
2. dementia, substance abuse etc. and other conditions seriously affecting cognitive and communication skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: approximately 1500 Chinese PDN outpatient patients were required
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
prevalnce of irrational use of pain reliever drugs | baseline
  percent

SECONDARY OUTCOMES:
Douleur Neuropathique4 questions(DN4) | baseline
  unit
Visual Analogue Score(VAS) | baseline
  1 to 10 units are minimum to maximum scores. Higher values represent a worse outcome of pain.
Patient Health Questionnaire(PHQ-9) | baseline
  0 to 27 units are minimum to maximum scores. Higher values represent a worse outcome of depression.
Generalized Anxiety Disorder Screener (GAD-7) | baseline
  0 to 21 units are minimum to maximum scores. Higher values represent a worse outcome of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Dongsheng Fan, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang Y, Zhang S, Pan L, Wang B, Sun Y, Gao L, Wang L, Cui L, Zhang Q, Shang H, Jin S, Qin X, Geng D, Yu X, Yang L, Li L, Li Z, Yan C, Sun H, Sun T, Du B, Cao J, Hu F, Ma J, Zhou S, Zhao F, Li W, Zheng J, Yi Y, Xu J, Hu B, Sheng B, Li Z, Zhao Z, Yang T, Wang N, Zhao H, Mima D, Qu H, Wang Y, Song F, Li X, Li N, Fan D. Painful Diabetic Peripheral Neuropathy Study of Chinese Outpatients (PDNSCOPE): A Multicentre Cross-Sectional Registry Study of Clinical Characteristics and Treatment in Mainland China. Pain Ther. 2021 Dec;10(2):1355-1373. doi: 10.1007/s40122-021-00281-w. Epub 2021 Aug 7. PMID 34363598
- [Derived] Zhang Y, Li N, Zhao Y, Fan D. Painful Diabetic Peripheral Neuropathy Study of Chinese OutPatiEnts (PDN-SCOPE): protocol for a multicentre cross-sectional registry study of clinical characteristics and treatment in China. BMJ Open. 2019 Apr 8;9(4):e025722. doi: 10.1136/bmjopen-2018-025722. PMID 30962233